CLINICAL TRIAL: NCT07066358
Title: Simultaneous Bilateral Radiofrequency Thalamotomy for Medication-Refractory Essential Tremor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo Women's Medical University (Other)
Responsible Party: Principal Investigator, Shiro Horisawa, Assistant Professor, Department of Neurosurgery, Tokyo Women's Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TWMU-Vim01
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Essential Tremor
Keywords: thalamotomy; intraoperative MRI
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: All enrolled participants will receive simultaneous bilateral radiofrequency lesioning of the ventral intermediate nucleus (Vim) of the thalamus in a single surgical session. No control or comparator group is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral RF Thalamotomy (Experimental): Participants in this arm will undergo simultaneous bilateral radiofrequency lesioning of the ventral intermediate nucleus (Vim) of the thalamus using a stereotactic frame under local anesthesia. The procedure begins with treatment on the side contralateral to the dominant hand. Intraoperative MRI will be performed after the first lesion to confirm the absence of hemorrhagic complications. If no complications are observed, the procedure will continue on the opposite side. If hemorrhage is detected, the surgery will be terminated after unilateral treatment. The goal of this intervention is to reduce medication-refractory tremor in both upper limbs.
  Interventions: Procedure: Simultaneous Bilateral RF Thalamotomy

INTERVENTIONS:
Procedure: Simultaneous Bilateral RF Thalamotomy — This intervention involves simultaneous bilateral radiofrequency (RF) lesioning of the ventral intermediate nucleus (Vim) of the thalamus using a stereotactic frame under local anesthesia. The procedure begins with RF ablation on the side contralateral to the dominant hand. Intraoperative MRI is then performed to confirm the absence of hemorrhagic complications. If no bleeding or other adverse events are detected, the procedure proceeds to the contralateral Vim. If hemorrhage is identified, the surgery is terminated after unilateral treatment. This technique allows for immediate bilateral tremor reduction in patients with medication-refractory essential tremor, while prioritizing patient safety through intraoperative imaging-based decision-making.

SUMMARY:
This study aims to evaluate the safety and effectiveness of simultaneous bilateral radiofrequency thalamotomy for patients with medication-refractory essential tremor (ET). Essential tremor is a common neurological condition that causes involuntary shaking, often affecting the hands and interfering with daily activities such as writing, eating, or using tools. While medications such as propranolol and primidone can help some patients, others experience limited or no benefit.

In this study, five adult participants diagnosed with essential tremor that does not respond to standard medications will undergo simultaneous bilateral stereotactic radiofrequency lesioning of the ventral intermediate nucleus (Vim) of the thalamus. This procedure involves precisely targeting both sides of the Vim to reduce tremor in both arms during a single surgical session.

Prior to surgery, participants will undergo brain MRI for surgical planning, as well as clinical evaluations including the Clinical Rating Scale for Tremor (CRST), Quality of Life in Essential Tremor Questionnaire (QUEST), the Scale for the Assessment and Rating of Ataxia (SARA), mood scales (BDI, BAI, AES), and cognitive function testing.

The surgery will be performed under local anesthesia using a stereotactic frame and intraoperative imaging. Tremor reduction will be assessed postoperatively and at 1, 3, and 6 months. The primary outcome is the improvement in CRST scores at 6 months. Secondary outcomes include quality of life (QUEST), ataxia symptoms (SARA), mood and cognitive changes, and adverse events.

This research is being conducted at Tokyo Women's Medical University. The study is IRB-approved and participants will be monitored closely throughout the 6-month follow-up period. Any complications or adverse events, such as temporary speech or swallowing difficulties, will be recorded and managed appropriately. The goal of this study is to explore whether performing thalamotomy on both sides simultaneously is a safe and effective treatment option for patients with severe and medication-resistant essential tremor.

DETAILED DESCRIPTION:
Essential tremor (ET) is one of the most common movement disorders, characterized by kinetic and postural tremor, particularly of the upper limbs. While the pathophysiology of ET is not fully understood, the ventral intermediate nucleus (Vim) of the thalamus plays a key role as a relay center in the tremor-generating network, making it a validated target for surgical interventions. Although unilateral thalamotomy has long been recognized as an effective treatment for drug-refractory ET, bilateral procedures have been limited due to concerns regarding adverse effects, particularly speech disturbance, dysphagia, and gait imbalance.

Recently, staged bilateral thalamotomies, especially using magnetic resonance-guided focused ultrasound (MRgFUS), have shown promising results. However, simultaneous bilateral thalamotomy using radiofrequency lesioning has rarely been systematically evaluated. Given the shorter surgical burden and potential for immediate bilateral tremor suppression, simultaneous bilateral thalamotomy may represent a meaningful therapeutic option in selected patients with severe, symmetrical, medication-resistant tremor.

This investigator-initiated, prospective, single-arm clinical trial is designed to evaluate the feasibility, safety, and efficacy of simultaneous bilateral radiofrequency thalamotomy targeting the Vim in patients with medication-refractory essential tremor. A total of five participants will be enrolled and undergo stereotactic lesioning in a single operative session.

Preoperative evaluations include structural brain MRI, Clinical Rating Scale for Tremor (CRST), Quality of Life in Essential Tremor Questionnaire (QUEST), Scale for the Assessment and Rating of Ataxia (SARA), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Apathy Evaluation Scale (AES), and Mini-Mental State Examination (MMSE). Surgical planning is based on direct targeting of the Vim using high-resolution MRI. The procedure will be performed under local anesthesia, with frame-based stereotactic guidance, and intraoperative CT or MRI will be used to monitor safety.

Lesioning will begin on the side contralateral to the dominant hand. After completing the first side, intraoperative MRI will be performed to confirm the absence of hemorrhagic complications. Only if no bleeding is detected will the procedure proceed to the contralateral Vim. If hemorrhage or other significant adverse events are identified after the first lesion, the surgery will be terminated after unilateral treatment. If no adverse events are found, lesioning will continue on the second side. The expected lesioning time is approximately 30 minutes per side. Postoperative imaging will be performed immediately after the procedure and the following day.

Postoperative assessments will be performed at discharge, and at 1 month, 3 months, and 6 months. CRST will be evaluated at each follow-up point, while QUEST and SARA will be repeated at 1, 3, and 6 months. Mood scales and MMSE will be reassessed at 6 months. MRI will also be repeated at 3 months to evaluate lesion location and any potential structural changes. The primary endpoint is the change in CRST score at 6 months postoperatively. Secondary endpoints include quality of life, cerebellar symptoms, adverse events, and neuropsychiatric effects.

Participants will be closely monitored for adverse events, including intracranial hemorrhage, dysarthria, dysphagia, numbness, ataxia, or other neurological complications. The expected adverse event rates are based on prior publications and include transient dysarthria (~10%), swallowing difficulties (~5%), and mild sensory symptoms (~5%). Serious adverse events such as hemorrhage are considered rare (<1%).

This study is approved by the Institutional Review Board of Tokyo Women's Medical University and adheres to the ethical principles outlined in the Declaration of Helsinki and Japan's Clinical Research Act. Written informed consent will be obtained from all participants prior to enrollment.

The findings from this study are expected to contribute to the evidence base for bilateral surgical treatment of essential tremor and may help to define the role of simultaneous bilateral Vim thalamotomy in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 70 years.
* Diagnosis of essential tremor by a neurologist or neurosurgeon specializing in movement disorders.
* Refractory to standard pharmacological therapy (e.g., propranolol, primidone, benzodiazepines, or alprenolol).
* Mini-Mental State Examination (MMSE) score ≥ 27.
* Able to undergo MRI.
* Provided written informed consent for participation in the study.

Exclusion Criteria:

* History or evidence of bleeding tendency.
* MRI contraindications (e.g., metallic implants, severe claustrophobia).
* Presence of intracranial pathology on preoperative MRI that would interfere with surgery.
* Pregnant or breastfeeding individuals.
* Any other condition that the principal investigator deems inappropriate for study participation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Rating Scale for Tremor (CRST) Score From Baseline to 6 Months Postoperatively | Baseline and 6 Months After Surgery
  The Clinical Rating Scale for Tremor (CRST) is a standardized scale used to evaluate tremor severity and its impact on motor function and activities of daily living. The total CRST score includes postural and action tremor, writing, pouring tasks, and disability ratings. Higher scores indicate greater severity. The primary outcome is the change in total CRST score from preoperative baseline to 6 months after the bilateral radiofrequency thalamotomy.

SECONDARY OUTCOMES:
Change in QUEST Score From Baseline to 6 Months Postoperatively | Baseline, 1 Month, 3 Months, and 6 Months After Surgery
  The Quality of Life in Essential Tremor Questionnaire (QUEST) is a disease-specific instrument used to assess the impact of essential tremor on patients' quality of life. It includes items related to physical, psychosocial, and communication aspects. Higher scores indicate greater impairment.
Change in SARA Score From Baseline to 6 Months Postoperatively | Baseline, 1 Month, 3 Months, and 6 Months After Surgery
  The Scale for the Assessment and Rating of Ataxia (SARA) is a clinical scale that measures cerebellar ataxia symptoms such as gait, stance, limb coordination, and speech. Scores range from 0 (no ataxia) to 40 (severe ataxia). Higher scores indicate more severe impairment.
Change in BDI Score From Baseline to 6 Months Postoperatively | Baseline and 6 Months After Surgery
  The Beck Depression Inventory (BDI) is a widely used 21-item self-report questionnaire for assessing the severity of depressive symptoms. Scores range from 0 to 63, with higher scores indicating more severe depression.
Change in BAI Score From Baseline to 6 Months Postoperatively | Baseline and 6 Months After Surgery
  The Beck Anxiety Inventory (BAI) is a 21-item self-report instrument used to assess the severity of anxiety symptoms in adults. Total scores range from 0 to 63, with higher scores reflecting greater anxiety.
Change in AES Score From Baseline to 6 Months Postoperatively | Baseline and 6 Months After Surgery
  The Apathy Evaluation Scale (AES) measures apathy in behavioral, cognitive, and emotional domains. It is a validated tool for assessing motivation and initiative, particularly in neurological populations. Higher scores indicate more severe apathy.

CONTACTS AND LOCATIONS:
Overall Officials: Shiro HORISAWA, MD, Principal Investigator — Tokyo Women's Medical University
Locations (1):
- Tokyo Women's Medical University, Department of Neurosurgery, Shinjuku-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data including clinical rating scales (e.g., QUEST, SARA, BDI, BAI, AES) will be shared. No personally identifiable information will be included.
Supporting Information: Study Protocol
Time Frame: The data will be available beginning 6 months after publication of the study results in a peer-reviewed journal and will be available for 5 years.
Access Criteria: Qualified researchers may request access to the de-identified individual participant data and supporting documents (Study Protocol, SAP, ICF). Access will be granted after approval by the principal investigator and a data use agreement.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT07066358/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT07066358/ICF_001.pdf